CLINICAL TRIAL: NCT04898673
Title: A Pre-Marketing, Prospective, Multi-Site, Open-Label, Within-Subject, Feasibility, Interventional Study of Speech Perception With Experienced Adult Cochlear Implant Recipients Using the CP1110 Sound Processor and Compared With the CP1000 Sound Processor
Brief Title: CP1110 Sound Processor Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5804
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-02

CONDITIONS: Adult Cochlear Implant Recipients

STUDY DESIGN:
Intervention Model Description: prospective, pre-market, Multi-site, non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CP1000 Sound Processor followed by the CP1110 Sound Processor (Experimental): All study subjects were provided with a unique identifier. The ones that ended in an odd number were administered the CP1000 Sound Processor followed by the CP1110 Sound Processor.
  Interventions: Device: CP1110; Device: CP1000
- CP1110 Sound Processor followed by the CP1000 Sound Processor (Experimental): All study subjects were provided with a unique identifier. The ones that ended in an even number were administered the CP1110 Sound Processor followed by the CP1000 Sound Processor.
  Interventions: Device: CP1110; Device: CP1000

INTERVENTIONS:
Device: CP1110 — Sound Processor
Device: CP1000 — Sound Processor

SUMMARY:
The clinical study aims to investigate the speech performance with the CP1110 Sound Processor, compared with the CP1000 Sound Processor, and inclusion of a noise reduction feature in the Automatic Scene Classifier..

DETAILED DESCRIPTION:
The study will build on the evidence previously collected on behind-the-ear sound processors and noise reduction, with particular focus on the speech perception performance of the CP1110 Sound Processor when compared to the CP1000 Sound Processor.

To assess the primary and secondary speech perception objectives, the study incorporates a within-subject repeated-measures design in which each subject will undergo in-booth speech perception testing with all combinations of hardware and signal processing settings in a sound booth. The average difference scores will indicate the performance difference for each of the paired comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Post lingually deafened
3. Implanted with the CI600 Series (CI612, CI632, CI622, CI624), CI500 Series (CI512, CI532, CI522) or Freedom Series (CI24RE(CA), CI24RE(ST), CI422)
4. At least 6 months experience with a cochlear implant.
5. At least 3 months experience with a Nucleus 6 (CP910/920), Kanso (CP950), Kanso 2 (CP1150) or Nucleus 7 (CP1000) Sound Processor
6. Able to score 30% or more at +15 SNR with CI alone on a sentence in babble test
7. Willingness to participate in and to comply with all requirements of the protocol.
8. Fluent speaker in English as determined by the investigator
9. Willing and able to provide written informed consent

Exclusion Criteria:

1. Additional disabilities that would prevent participation in evaluations.
2. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedures.
3. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
4. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
5. Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
6. Currently participating, or participated in another interventional clinical study/trial in the past 30 days, or (if less than 30 days) the prior investigation was Cochlear sponsored and determined by the investigator to not impact clinical findings of this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cochlear Sydney, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 subjects were recruited.
Period: Overall Study
Arm/Group | CP1000 Sound Processor Followed by the CP1110 Sound Processor | CP1110 Sound Processor Followed by the CP1000 Sound Processor
Started | 11 | 10
CP1110 Sound Processor | 10 | 10
CP1000 Sound Processor | 10 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Screenfail | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Baseline characteristics are combined across the 2 arms.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Customized [Median (Full Range); unit: years] | 64.5 [33.0 to 91.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 20

OUTCOME MEASURES:

1. Primary Outcome: Speech Reception Thresholds (SRT) Assessed Via Sentence Scores in Spatially Separated Adaptive Noise
Description: Paired difference in dB SRT between treatment and control, with their applicable noise reduction feature enabled.
  The speech recognition threshold (SRT) examines at which level the participant can repeat 50% of the speech material correctly. These scores may be negative or positive numeric values. Lower dB SRT scores indicate a better outcome.
Time Frame: One day
Measure: Mean (95% Confidence Interval); unit: decibels
Groups:
- CP1000: All subjects tested using CP1000
- CP1110: All subjects tested using CP1110
Arm/Group | CP1000 | CP1110
Number analyzed (Participants) | 20 | 20
decibels | -6.07 [-6.07 to -4.47] | -11.30 [-13.28 to -9.32]
Statistical Analysis 1: Comparison: CP1000 vs CP1110; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = -5.23, 95% CI 2-sided [-6.08 to -4.37], Standard Error of Mean 0.41

2. Secondary Outcome: Percentage of Correct Words Assessed by CNC (Consonant Nucleus Consonant) Monosyllabic Word Scores in Quiet
Description: Paired differences in percentage CNC Words correct in quiet (50 dB) between treatment and control, with various configurations of signal processing settings being enabled or disabled for each measure. Word recognition is a score of the number of words correctly repeated, expressed as a percentage. Higher percentage scores indicate a better outcome.
  Secondary Endpoint 1: CNC Words correct in quiet (50 dB) with both CP1000 and CP1110 sound processors using Signal-to-Noise Ratio - Noise Reduction (SNR-NR) turned on.
Time Frame: One day
Measure: Mean (95% Confidence Interval); unit: percentage of correct words
Arm/Group | CP1000 | CP1110
Number analyzed (Participants) | 20 | 20
percentage of correct words | 57.5 [51.67 to 63.33] | 58.10 [51.56 to 64.64]
Statistical Analysis 1: Comparison: CP1000 vs CP1110; Test type: Superiority; p = 0.670, ANOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.31 to 3.51], Standard Error of Mean 1.39

3. Secondary Outcome: Percentage of Correct Assessed by CNC (Consonant Nucleus Consonant) Monosyllabic Word Scores in Quiet
Description: Paired differences in percentage CNC Words correct in quiet (50 dB) between treatment and control, with various configurations of signal processing settings being enabled or disabled for each measure. Word recognition is a score of the number of words correctly repeated, expressed as a percentage. Higher percentage scores indicate a better outcome.
  CNC Words in Quiet Score using both CP1110 and CP1000 sound processors Signal-to-Noise Ratio - Noise Reduction (SNR-NR) off with expander on.
Time Frame: One day
Measure: Mean (95% Confidence Interval); unit: percentage of correct words
Groups:
- CP1000: All subjects tested with CP1000
- CP1110: All subjects tested with CP1110
Arm/Group | CP1000 | CP1110
Number analyzed (Participants) | 20 | 20
percentage of correct words | 60.90 [54.98 to 66.82] | 57.15 [50.26 to 64.04]
Statistical Analysis 1: Comparison: CP1000 vs CP1110; Test type: Non-Inferiority — Non-inferiority margin=-10% words correct; CP1110 non-inferior to CP1000 if the lower limit of the confidence interval for the difference > -10% words correct; p = 0.026, ANOVA; Mean Difference (Final Values) = -3.75, 95% CI 2-sided [-7.00 to -0.50], Standard Error of Mean 1.55

4. Secondary Outcome: Percentage of Correct Words Assessed by CNC (Consonant Nucleus Consonant) Monosyllabic Word Scores in Quiet
Description: Paired differences in percentage CNC Words correct in quiet (50 dB) between treatment and control, with various configurations of signal processing settings being enabled or disabled for each measure.
  Word recognition is a score of the number of words correctly repeated, expressed as a percentage. Higher percentage scores indicate a better outcome.
  CNC Words in Quiet Score of CP1110 sound processor ForwardFocus ON (Moderate) vs CP1000 sound processor Signal-to-Noise Ration-Noise Reduction) On.
Time Frame: One Day
Measure: Mean (95% Confidence Interval); unit: percentage of correct words
Arm/Group | CP1000 | CP1110
Number analyzed (Participants) | 20 | 20
percentage of correct words | 57.50 [51.67 to 63.33] | 56.35 [50.33 to 62.37]
Statistical Analysis 1: Comparison: CP1000 vs CP1110; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.411, ANOVA; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-4.02 to 1.72], Standard Error of Mean 1.37

ADVERSE EVENTS:
Time Frame: 2 months
Description: All study subjects were provided with a unique identifier .The ones that ended in an odd number were administered the CP1000 Sound Processor followed by the CP1110 Sound Processor, and the opposite order was used for participants with an even numbered subject identifier.
Groups:
- CP1000 Sound Processor: All study participants whilst using CP1000 Sound Processor
- CP1110 Sound Processor: All study participants whilst using CP1110 Sound Processor
Arm/Group | CP1000 Sound Processor | CP1110 Sound Processor
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT04898673/Prot_002.pdf
  • Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT04898673/SAP_001.pdf